CLINICAL TRIAL: NCT04581785
Title: A Phase 1/2 Open-label Clinical Study of hLB-001 Gene Therapy in Pediatric Patients With Methylmalonic Acidemia Characterized by MMUT Mutations
Brief Title: Gene Therapy With hLB-001 in Pediatric Patients With Severe Methylmalonic Acidemia
Acronym: SUNRISE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to low likelihood of clinical benefit in treated participants.
Sponsor: LogicBio Therapeutics, Inc (Industry)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB001-001
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Methylmalonic Acidemia
Keywords: inborn errors of metabolism; mut0; mut-; mut deficiency; organic acidemia; SUNRISE
MeSH Terms: conditions — Methylmalonic acidemia; Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 1 Part A (Experimental): 3 year-olds to 12 year-olds
  Interventions: Biological: hLB-001
- Dose Level 1 Part B (Experimental): 6 month to 2 year-olds
  Interventions: Biological: hLB-001
- Dose Level 1 Part C (Experimental): 6 month to 12 year-olds
  Interventions: Biological: hLB-001
- Dose Level 2 Part A (Experimental): 3 year-olds to 12 year-olds
  Interventions: Biological: hLB-001
- Dose Level 2 Part B (Experimental): 6 month to 2 year-olds
  Interventions: Biological: hLB-001

INTERVENTIONS:
Biological: hLB-001 — hLB-001 via IV infusion

SUMMARY:
The SUNRISE trial is a first-in-human (FIH), open-label, Phase 1/2 clinical trial designed to assess the safety, tolerability and preliminary efficacy of a single intravenous infusion of hLB-001 in pediatric patients with MMA characterized by methylmalonyl-CoA mutase gene (MMUT) mutations. hLB-001 is a liver-targeted, recombinant engineered adeno-associated viral (rAAV) vector utilizing the LK03 capsid (rAAV-LK03), designed to non-disruptively integrate the human methylmalonyl-CoA mutase gene at the albumin locus.

The trial is expected to enroll pediatric patients with ages ranging from 6 months to 12 years, initially starting with 3 to 12 year-old patients and then adding patients aged 6 months to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* At the time of dosing, participants must be 6 months to 12 years of age
* Males and females with diagnosis of severe MMA meeting all the following;

  1. Isolated MMA with genetically confirmed, pathogenic mutations in the MMUT gene
  2. Screening serum/plasma methylmalonic acid level of >100 µmol/L
  3. One or more of the following considered by the PI to be MMA-related: (i) An unscheduled ER visit, hospitalization or requirement for sick day diet in the year prior to screening visit (ii) Developmental delay, movement disorder, optic neuropathy or feeding disorder with tube feeding requirement
  4. Medically stable for the 2 months prior to the start of screening

Exclusion Criteria:

* Participants with organic acidemias other than isolated MMA, or with any other causes of hyperammonemia
* Having received MMA-targeted gene therapy or nucleic acid therapy
* Participants on insulin or high dose hydroxocobalamin (> 1 mg/day OHB12 parenteral)
* Kidney or liver transplant, including hepatocyte cell therapy
* Estimated glomerular filtration rate (eGFR) of < 60 mL/min/1.73 m2 based on age appropriate equations, or ongoing dialysis for renal disease
* Participant tests positive for anti-rAAV-LK03-neutralizing antibodies

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=LB001-001&attachmentIdentifier=9b2b0d4e-d9d4-4487-929e-b59ffa9dc33e&fileName=LogicBio_LB001_001_abbrev_CSR_Synopsis_final_07FEB24_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to enroll participants in 2 Cohorts. Cohort 1 consisted of 2 parts: Part A enrolled participants aged 3 to 12 years, and Part B enrolled participants aged 6 months to 36 months. Part C was to enroll participants aged 6 months to 12 years for further safety evaluation prior to enrolling participants in Cohort 2. No participants were enrolled in Part C and thus Cohort 2 was not initiated.
Groups:
- Cohort 1 Part A: 3- to 12-years Old: Participants 3- to 12-years old received a single intravenous (IV) infusion of hLB-001.
- Cohort 1 Part B: 6- to 36-months Old: Participants 6- to 36-months old received a single IV infusion of hLB-001.
Period: Overall Study
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Started | 2 | 2
Received at Least 1 Dose of Study Drug | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug. Cohorts have been combined in the Baseline Characteristics section to maintain participant confidentiality.
Groups:
- Overall Participants (Cohort 1 Part A and Part B): Participants received a single IV infusion of hLB-001.
Arm/Group | Overall Participants (Cohort 1 Part A and Part B)
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: months] | 48.5 [20 to 113]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAE was an AE that was not present prior to administration of hLB-001, or an event already present that worsened in either severity or frequency following hLB-001administration. A summary of serious adverse events (SAEs) and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: From first dose of study drug up to Week 52
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 Part A: 3- to 12-years Old: Participants 3- to 12-years old received a single IV infusion of hLB-001.
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Number of Participants With Infusional Toxicities
Description: An infusional toxicity was a hLB-001-related AE that limits, delays, or requires medical intervention during administration. A summary of SAEs and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline up to Week 52
Population: The safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

3. Secondary Outcome: Change From Baseline in Serum Methylmalonic Acid Level at Week 52
Time Frame: Baseline, Week 52
Population: The intent-to-treat (ITT) population included all participants receiving hLB-001 who had baseline data and at least 1 postdose measurement.
Measure: Median (Full Range); unit: micromoles (µmol)/liter (L)
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
micromoles (µmol)/liter (L) | 286.90 [256.1 to 317.7] | 122.72 [116.0 to 129.5]

4. Secondary Outcome: Change From Baseline in Serum Methylcitrate Level at Week 52
Time Frame: Baseline, Week 52
Population: The ITT population included all participants receiving hLB-001 who had baseline data and at least 1 postdose measurement.
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
µmol/L | 2.35 [1.5 to 3.2] | 4.66 [4.4 to 4.9]

5. Secondary Outcome: Change From Baseline in Serum Fibroblast Growth Factor 21 (FGF21) Level at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
µmol/L | -4.75 [-7.6 to -1.9] | 1.57 [0.7 to 2.4]

6. Secondary Outcome: Percent Change From Baseline in Propionate Oxidation Rate at Week 52
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
percent change | 6.28 [5.2 to 7.3] | 2.16 [1.6 to 2.8]

7. Secondary Outcome: Change From Baseline in Serum Albumin-2A Level at Week 52
Description: Below the limit of quantification (BLQ) value was 2.44 nanograms (ng)/milliliter (mL).
Time Frame: Baseline, Week 52
Population: as for outcome 4
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
Number analyzed (Participants) | 2 | 2
µmol/L | NA [NA to NA] — NA=Not available. Insufficient data above BLQ available for this Outcome Measure. | NA [NA to NA] — NA=Not available. Insufficient data above BLQ available for this Outcome Measure.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 52
Description: The safety population included all participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1 Part A: 3- to 12-years Old | Cohort 1 Part B: 6- to 36-months Old
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Part A: 3- to 12-years Old (N=2) | Cohort 1 Part B: 6- to 36-months Old (N=2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Part A: 3- to 12-years Old (N=2) | Cohort 1 Part B: 6- to 36-months Old (N=2)
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1
Transaminases increased (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low likelihood of clinical benefit in treated participants. Hence; no participants were enrolled in Part C and thus Cohort 2 was not initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT04581785/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT04581785/SAP_001.pdf